CLINICAL TRIAL: NCT03471949
Title: Evaluation of the Profile of Blood Glucose Using Dexcom G4 in a Population With Normal Oral Glucose Tolerance Test
Brief Title: Dexcom G4 in a Population With Normal Oral Glucose Tolerance Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CGM and healthy population
Record Dates: First submitted 2017-12-18; First posted 2018-03-21 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CGM in a population with normal OGTT (Experimental): A non-randomized, days 1-7 blinded, and days 8-14 non-blinded Dexcom G4 (CGM) trial. Each subject will sample capillary blood with the HemoCue meter and measure the concentration of glucose, minimum 3 times per day for 14 days.
  Interventions: Other: CGM in a population with normal OGTT

INTERVENTIONS:
Other: CGM in a population with normal OGTT — The population with normal OGTT will use CGM and document their values as well as be documenting a capillary blood glucose value

SUMMARY:
The purpose of this study was to obtain reference values of CGM in healthy individuals using the Dexcom G4 sensor and evaluate whether reported low glucose values by the Dexcom G4 sensor are really low when confirmed by capillary testing.

DETAILED DESCRIPTION:
Evaluation of the profile of blood glucose using Dexcom G4 in a population with normal oral glucose tolerance test. The investigators have used information from a previous study of 60 participants using Dexcom G4, CGM system. A non-randomized, days 1-7 blinded and days 8-14 non-blinded CGM trial, the study was performed to evaluate the profile of blood glucose using CGM in the population with normal oral glucose tolerance test (OGTT). All enrolled subjects with at least three time-points with evaluable values from CGM system and the reference capillary value obtained from HemoCue during the whole study period were included in the Intent-to-Treat (ITT) population

ELIGIBILITY:
Inclusion Criteria:

1. Normal oral glucose tolerance test
2. Normal HbA1c value
3. Age of 18 years or older

Exclusion Criteria:

1. Known diabetes
2. Known prediabetes
3. Corticosteroid use during the last month
4. Planned corticosteroid use during the study
5. Pregnancy or planned pregnancy during the study period
6. Paracetamol use during the last 2 days
7. Planned paracetamol use during the study
8. Allergy to any adhesives used for CGM or clorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
The percentage of time with low CGM values ( blood glucose <4.0 mmol/l) | Day 1-7
  Percentage of time with low CGM values, Measured by continuous glucose monitoring (CGM) (<72 mg/dL, <4.0 mmol/L) estimated on days 1-7 when participants used masked CGM.

SECONDARY OUTCOMES:
The percentage of time with low CGM values (blood glucose <3.0 mmol/l) | Day 1-7
  Measured by continuous glucose monitoring (CGM) and the percentage of time with low CGM values (<54 mg/dL, <3.0 mmol/L) evaluated on days 1-7
The difference in mean glucose levels between days 1-7 and day 8-14 | Day 1-7 and day 8-14
  Measured by continuous glucose monitoring (CGM) between day 1-7 and 8-14
The percentage of time with glucose levels in euglycaemic range (72-126 mg/dL) | Day 1-14
  Measured by continuous glucose monitoring (CGM) (72-126 mg/dL, 4-7 mmol/L) between day 1-7 and 8-14
The percentage of time with glucose levels in euglycaemic range (72-180 mg/dL) | Day 1-14
  Measured by continuous glucose monitoring (CGM) (72-180 mg/dL, 4-10 mmol/L) between day 1-7 and 8-14
The percentage of time with glucose levels in hyperglycaemic range (>198 mg/dL) | Day 1-14
  Measured by continuous glucose monitoring (CGM) with high glucose levels (>198 mg/dL, >11 mmol/L) between day 1-7 and 8-14
The percentage of time with glucose levels in hyperglycaemic range (>252 mg/dL) | Day 1-14
  Measured by continuous glucose monitoring (CGM) with high glucose (>252 mg/dL, >14 mmol/L) between day 1-7 and 8-14
The Standard Deviation (SD) | Day 1-7 and day 8-14
  Difference in standard deviation of glucose levels measured by CGM between day 1-7 and day 8-14
The evaluation of experience of the CGM, glucose monitoring systems. | Week 2, day14
  Evaluation of the Dexcom G4 system from questionnaire regarding the following questions, 1. The visual analogue scale 1-100 mm. How do you experience the benefits of seeing your daily blood glucose profile with the help of CGM (continuous glucose monitoring)? The evaluation of questions of the Dexcom G4 system were expressed on a 0-100 scale with lowest value (0) equaling to Not rewarding at all and highest value (100) equaling to completely rewarding.
  2. Do you consider the CGM can be a great educational tool for patients who are at risk for getting diabetes? (yes, no)
  3. Can CGM give you a mindset about diet and lifestyle changes? (yes, no)
  4. Can you describe your experiences using CGM?
Difference in Mean Amplitude of Glycemic Excursions (MAGE) | Day 1-7, Day 8-14
  Difference in mean amplitude glucose excursion (MAGE) measured by CGM between day 1-7 and 8-14
Mean Absolute Relative Difference (MARD) | Day 1-14
  Mean Absolute Relative Difference (MARD) estimated from HemoCue glucose values and CGM-values from days 1-14.
Mean Absolute Difference (MAD) | Day 1-7, Day 8-14
  Measured by continuous glucose monitoring (CGM) between day 1-7 and 8-14
Coefficient of Variation (CV) | Day 1-7, Day 8-14
  Difference in coefficient of variation measured by continuous glucose monitoring (CGM) between day 1-7 and 8-14
Pearson correlation coefficient | Day 8-14
  Pearson correlation coefficient estimated from HemoCue and CGM glucose values from days 8-14.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus MD Lind, Phd, Principal Investigator — Study Principal Investigator, Nu-Hospital Group, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sofizadeh S, Pehrsson A, Olafsdottir AF, Lind M. Evaluation of Reference Metrics for Continuous Glucose Monitoring in Persons Without Diabetes and Prediabetes. J Diabetes Sci Technol. 2022 Mar;16(2):373-382. doi: 10.1177/1932296820965599. Epub 2020 Oct 26. PMID 33100059